CLINICAL TRIAL: NCT01240135
Title: Clinical Performance of a Marketed Silicone Hydrogel Contact Lens When Used With Silicone Hydrogel MPDS FID 114675A
Brief Title: Clinical Performance of a Silicone Hydrogel Lens With Use of FID 114675A
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Supportive Care
Other Study IDs: C-10-030
Record Dates: First submitted 2010-11-10; First posted 2010-11-15 (Estimated); Results first posted 2012-07-12 (Estimated); Last update posted 2012-07-12 (Estimated); Status verified 2012-06

CONDITIONS: Contact Lens Fit; Myopia
Keywords: Contact Lens Wear; Contact Lens Solution; Multi-purpose disinfecting solution; Myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- FID 114576A / renu fresh (Other): FID 114675A used for contact lens care per protocol-specified instructions for 14 days, followed by a minimum 1-day washout period, after which renu fresh used for contact lens care for an additional 14 days.
  Interventions: Device: FID 114675A multi-purpose disinfecting solution (MPDS); Device: renu fresh Multi-Purpose Solution (MPS); Device: Galyfilcon A contact lenses (Acuvue Advance)
- renu fresh / FID 114675A (Other): Renu fresh used for contact lens care per protocol-specified instructions for 14 days, followed by a minimum 1-day washout period, after FID 114675A used for contact lens care for an additional 14 days.
  Interventions: Device: FID 114675A multi-purpose disinfecting solution (MPDS); Device: renu fresh Multi-Purpose Solution (MPS); Device: Galyfilcon A contact lenses (Acuvue Advance)

INTERVENTIONS:
Device: FID 114675A multi-purpose disinfecting solution (MPDS) — Daily regimen, 14 days: Thoroughly wet and rub each side of study contact lens for 10 seconds, rinse each side of the lens for 10 seconds, and soak contact lens for at least 6 hours.
  Other Names: Alcon Multi-Purpose Disinfecting Solution (MPDS)
Device: renu fresh Multi-Purpose Solution (MPS) — Daily regimen, 14 days: Wet study contact lens with 3 drops and rub each side of the lens for 20 seconds, rinse each side of the lens for 5 seconds, and soak contact lens for at least 4 hours.
  Other Names: Bausch + Lomb renu® fresh™ Multi-Purpose Solution
Device: Galyfilcon A contact lenses (Acuvue Advance) — A fresh pair of contact lenses matching subject's pre-study lenses, including parameters, dispensed at the beginning of each period for daily wear, minimum 8 hours per day, 14 days.
  Other Names: Acuvue® Advance®

SUMMARY:
The purpose of this study is to evaluate the clinical performance of a silicone hydrogel contact lens when used with an investigational multi-purpose disinfecting solution (MPDS).

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older.
* History of at least 5 days successful daily wear (minimum 8 hours per day) of spherical, single power Acuvue® Advance® SiH contact lenses prior to Visit 1.
* Wear contact lenses a minimum of 8 hours per day prior to Visit 1.
* Vision correctable to 20/30 (Snellen) or better in each eye at distance with study lenses at Visit 1.
* Other protocol-defined inclusion criteria may apply.

Exclusion Criteria:

* Need to wear contact lenses on an extended wear basis (i.e., overnight) during the study.
* Use of products other than a multi-purpose solution to care for lenses at least 7 days prior to Visit 1. Pre-study use of rewetting drops is acceptable.
* History of intolerance or known sensitivity to any component of the treatments.
* Use of over-the-counter (OTC) or prescribed topical ocular medications within 7 days prior to Visit 1.
* Other protocol-defined exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2010-10; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from 5 US study centers.
Period: Period One, 14 Days of Wear
Arm/Group | FID 114576A / Renu Fresh | Renu Fresh / FID 114675A
Started | 44 | 45
Completed | 44 | 45
Not Completed | 0 | 0
Period: Period Two, 14 Days of Wear
Arm/Group | FID 114576A / Renu Fresh | Renu Fresh / FID 114675A
Started | 44 | 45
Completed | 43 | 43
Not Completed | 1 | 2
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Adverse Event | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | FID 114576A / Renu Fresh | Renu Fresh / FID 114675A | Total
Number analyzed (Participants) | 44 | 45 | 89
Age Continuous [Mean (Standard Deviation); unit: years] | 34.3 (11.44) | 31.4 (9.71) | 32.8 (10.64)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 30 | 61
  Male | 13 | 15 | 28

OUTCOME MEASURES:

1. Primary Outcome: Lens Fit
Description: As assessed by the investigator using a composite score based on three lens fit measures: static, push-up, and centration. Static and pushup were assessed on a 5-point scale, where -2=reduced movement unacceptable, -1=reduced movement acceptable, 0=optimal movement, 1=excessive movement acceptable, 2=excessive movement unacceptable. Centration was assessed on a 3-point scale, where 0=optimal lens centration, 1=acceptable decentration, 2=unacceptable decentration. A subject with an assessment of optimal or acceptable for each measure was considered acceptable on all measurements.
Time Frame: Day 14 of lens wear
Population: Intent to treat: All randomized subjects with at least one post-baseline assessment after dispensing, according to randomized treatment.
Measure: Number; unit: percentage of acceptable fit
Groups:
- FID 114576A: FID 114675A used for contact lens care per protocol-specified instructions for 14 days.
- Renu Fresh: Renu fresh used for contact lens care per protocol-specified instructions for 14 days.
Arm/Group | FID 114576A | Renu Fresh
Number analyzed (Participants) | 87 | 88
percentage of acceptable fit | 100 | 100

2. Secondary Outcome: Mean Change From Baseline for Circumlimbal Conjunctival Staining Sum Score
Description: The bulbar conjunctiva was assessed by the investigator at baseline and Day 14 utilizing a slit-lamp and ophthalmic dye. Staining coverage was scored separately in each of four regions (nasal, temporal, inferior, and superior) using a 5-point photographic reference scale, where 0=0.00% coverage and 4=10% or greater coverage. The scores for the four regions were summed, with a sum score range of 0-16.
Time Frame: Day 14 of lens wear
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | FID 114576A | Renu Fresh
Number analyzed (Participants) | 87 | 88
units on a scale | 0.6 (2.49) | 1.4 (2.63)

ADVERSE EVENTS:
Time Frame: Adverse events were collected for the duration of the study: 11 October 2010 through 2 February 2011.
Description: All subjects who used study treatment or potentially used study treatment were evaluated for safety analysis.
Arm/Group | FID 114576A | Renu Fresh
Serious Adverse Events (participants affected / at risk) | 0/89 | 0/89
Other Adverse Events (participants affected / at risk) | 0/89 | 0/89

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Alcon reserves the right of prior review of any publication or presentation of information related to the study.